CLINICAL TRIAL: NCT04729634
Title: Survey Of Mobilisation and Breathing Exercises After Thoracic and Abdominal Surgery
Acronym: SOMBATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FoU i VGR: 275327
Record Dates: First submitted 2021-01-04; First posted 2021-01-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Abdominal Cancer; Heart Diseases
Keywords: Immobilization; Abdominal surgery; Thoracic surgery; Breathing training
MeSH Terms: conditions — Heart Diseases | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: A cohort of patients followed over time
Masking Description: The patients will not be aware of the study activities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobilization and breathing training (Other): Usual clinical care
  Interventions: Other: Mobilization

INTERVENTIONS:
Other: Mobilization — Mobilization and breathing exercises according to clinical care
  Other Names: Breathing training

SUMMARY:
Background

Thoracic or abdominal surgeries are followed by a shorter or longer period of immobilization and after major surgery there is a higher risk of developing cardiorespiratory complications. To prevent these complications, the patient is encouraged to change position and exercise in bed, get out of bed as early and as much as possible after the operation and to breathe with or without aids. There is no general definition of early mobilization and may start within a few hours to a few days after surgery. There is currently a lack of knowledge nationally and internationally about when the mobilization starts and what it contains.

Many patients also receive breathing training in connection with the surgery. There is currently no consensus on which method is preferable for which groups of patients. There are similarities and differences in practice in the world regarding postoperative breathing training. There are studies that have mapped practice after primarily thoracic surgery but also abdominal surgery. However, there are no studies that have mapped when the prescribed breathing training starts after different types of operations.

The purpose of the study is to map when mobilization and breathing training starts after abdominal and thoracic surgery and what is then performed

Method The study will be carried out as a quality follow-up with mapping of practice. Patients ≥ 18 years of age who are undergoing a planned or acute open, keyhole or robot-assisted surgery, who are extubated and who breathe spontaneously will be included. Exclusion criteria are completed plastic, trauma, orthopedic or transplant surgery.

The material will be recruited from Swedish university hospitals and county hospitals for 20 days of surgery (Monday through Thursday) for five consecutive weeks.

Clinical benefit The study will mean that clinical practice is presented which, with regard to mobilization, is the first study ever that will present when this takes place and what is done and, with regard to breathing training, the first that shows when this training is initiated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* undergoing a planned or acute open, laparoscopic or robot-assisted surgeon in the thorax or abdomen
* who are extubated within 24 h of surgery
* breathe spontaneously within 24 h of surgery

Exclusion Criteria:

* reconstructive-, trauma-, transplantation- or orthopedic surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1492 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
When mobilization starts after surgery | Within 24 hours after surgery
  Time from termination of anaesthesia to when mobilization starts, ie when the patients are sitting with the legs over the edge of the bed
Mobilization- Content | Within 24 hours after surgery
  Content of the mobilization performed i.e. which level of mobilization (sitting on the edge of the bed, standing by the bed, sitting in a chair and walking) which is reached.
Mobilization- Duration | Within 24 hours after surgery
  Duration of the mobilization performed, minutes
When any intervention with breathing exercises starts after surgery | Within 24 hours after surgery
  Time from termination of anesthesia to when the breathing exercise starts
Breathing exercise- Content | Within 24 hours after surgery
  Type of breathing exercise, as deep breathing, positive expiratory pressure or incentive spirometry.
Breathing exercise- Intensity | Within 24 hours after surgery
  Intensity of breathing exercise prescribed, sessions/time.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Fagevik Olsen M, Svensson-Raskh A, Westerdahl E, Nygren Bonnier M, Reeve J, Sehlin M. Current practice of targeted breathing exercises after abdominal and cardiothoracic surgery: a national multicentre observational study. Physiotherapy. 2025 Jun;127:101462. doi: 10.1016/j.physio.2024.101462. Epub 2024 Dec 24. PMID 39946932
- [Derived] Westerdahl E, Lilliecrona J, Sehlin M, Svensson-Raskh A, Nygren-Bonnier M, Olsen MF. First initiation of mobilization out of bed after cardiac surgery - an observational cross-sectional study in Sweden. J Cardiothorac Surg. 2024 Jul 4;19(1):420. doi: 10.1186/s13019-024-02915-4. PMID 38961385
- [Derived] Fagevik Olsen M, Sehlin M, Westerdahl E, Schandl A, Block L, Nygren-Bonnier M, Svensson-Raskh A. First mobilisation after abdominal and cardiothoracic surgery: when is it actually performed? A national, multicentre, cross-sectional study. BMJ Open. 2024 Feb 29;14(2):e082239. doi: 10.1136/bmjopen-2023-082239. PMID 38423778